CLINICAL TRIAL: NCT04075786
Title: Survey of Dysmorphic Uterus Knowledge Among Gynecologists.
Acronym: DUS-1
Status: Not yet recruiting | Type: Observational
Sponsor: Università degli Studi dell'Insubria (Other)
Collaborators: University of Miami (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, Università degli Studi dell'Insubria
Other Study IDs: Dysmorphic Uterus Survey-1
Record Dates: First submitted 2019-08-26; First posted 2019-09-03 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Dysmorphic Uterus
Keywords: Uterine malformations; Hysteroscopy; 3D ultrasound; Infertility
MeSH Terms: conditions — Uterine Anomalies; Infertility | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gynecologists: Gynecologists in active clinical practice and resident (in training) gynecologists.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Each participant will be shown 40 (forty) 3D ultrasound images of uterus of normal women without infertility and 40 (forty) infertile women with uterus with narrowing in the middle third diagnosed by hysteroscopy + 3D ultrasound and associated infertility (T, Y or I shaped).

SUMMARY:
Uterine malformations were initially described by Cruveilhier and Von Rokitansky in the 1800s. Many proposed classifications had been presented over the years, although only two are mostly used worldwide: the first proposed by the American Fertility Society (AFS) and the one recently published by European Society on Gynecologic Endoscopy / European Society of Human Reproductive Endocrinology (ESGE/ESHRE). Both classifications describe a special type of uterus, with an abnormally shaped narrow uterine cavity. This type of uterus was initially defined, before the use of ultrasound, as "hypoplasic uterus" by K. Menge and K.V. Oettingen in 1930. Subsequently, the AFS in its classification defined it as type VII as Diethylstilbestrol-related and the ESGE/ESHRE classification defined it as class U1a or T-shaped uterus.

At present there are no clear diagnostic criteria for this type of uterus and the only parameter widely accepted is that of "narrow uterine cavity due to thickened lateral walls". The purpose of this study is to conduct a survey of gynecologists in active clinical practice and resident (in training) gynecologists to establish the degree of concordance when cataloging 3D ultrasound images of normal or dysmorphic uteri, with the aim to identify common parameters that allow to identify the dysmorphic uterus with narrowing of the side walls.

The study will be carried out in two stages: in an initial step, participants will complete a survey evaluating their knowledge of uterine malformations and their involvement in assisted reproduction in their current clinical practice.

In the second step, participants will then watch a video of hysteroscopies and 3D ultrasound images of different cases highlighting the hysteroscopic/ultrasound correlation of the different variants of the uterus with narrowing of the side walls. Each participant will be shown 40 (forty) 3D ultrasound images of uterus of normal women without infertility and 40 (forty) infertile women with uterus with narrowing in the middle third diagnosed by hysteroscopy + 3D ultrasound and associated infertility (in T, Y or I shape). Once the survey is finished, the degree of concordance will be evaluated, with the aim to identify common parameters of diagnosis of dysmorphic uterus by 3D ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Practicing gynecologist specialist or fellow/resident (in training);
* Knowledge of the ESGE/AFS and T-Y-I uterine anomalies classification.

Exclusion Criteria:

• None.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Gynecologists in active clinical practice and resident (in training) gynecologists
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Degree of concordance between anticipated and actual diagnosis of dysmorphic uteri | Through study completion, an average of 1 year
  Degree of concordance will be expressed as the percentage of the investigated population that will identify correctly the diagnosis of dysmorphic uteri, distinguishing them from normal-shaped uteri, looking at the images obtained by ultrasound and hysteroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carugno, M.D., Study Director — University of Miami; Luis Alonso, M.D., Study Director — Centro Gutenberg, Malaga; Antonio Simone Laganà, M.D., Study Chair — Università degli Studi dell'Insubria

IPD SHARING:
Plan to Share IPD: Undecided